CLINICAL TRIAL: NCT01572909
Title: A Phase 2a Trial to Evaluate the Safety, Tolerability and Efficacy of Intravenous MTP-131 on Reperfusion Injury in Patients Undergoing Primary Percutaneous Coronary Intervention and Stenting for ST-segment Elevation Myocardial Infarction Infarction
Brief Title: Evaluation of Myocardial Effects of MTP-131 for Reducing Reperfusion Injury in Patients With Acute Coronary Events
Acronym: EMBRACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPIRI-201
Record Dates: First submitted 2012-03-28; First posted 2012-04-06 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Reperfusion Injury; STEMI
Keywords: Myocardial Reperfusion; Primary PCI; Stenting for ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — Reperfusion Injury; ST Elevation Myocardial Infarction | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendavia™ (Active Comparator): Bendavia™ administered intravenously at 0.05 mg/kg/hr at least 15, but no more than 60 minutes, prior to the anticipated time of the PCI, and continued for 1 hour after re-establishment of blood flow through the culprit vessel.
  Interventions: Drug: Bendavia (MTP-131)
- Placebo (Placebo Comparator): Placebo administered intravenously at 60 mL/hr at least 15, but no more than 60 minutes, prior to the anticipated time of the PCI, and continued for 1 hour after re-establishment of blood flow through the culprit vessel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bendavia (MTP-131) — 0.05 mg/kg/hr
  Other Names: MTP-131; Elamipretide
  Arms: Bendavia™
Drug: Placebo — Identically appearing placebo
  Arms: Placebo

SUMMARY:
The EMBRACE-STEMI trial was a Phase 2a prospective, multicenter, multinational randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, and efficacy of IV administered elamipretide (also known as MTP-131, or Bendavia) on a background of standard-of-care therapy for reduction of reperfusion injury in patients with first time acute, anterior wall ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
The EMBRACE-STEMI trial was a Phase 2a prospective, multicenter, multinational randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, and efficacy of IV administered elamipretide on a background of standard-of-care therapy for reduction of reperfusion injury in patients with first time acute, anterior wall STEMI.

Patients were randomized to receive either an infusion of elamipretide at 0.05 mg/kg/hr or an identically appearing placebo administered as an IV infusion at 60 mL/hr. The infusion began at least 15 minutes but no more than 1 hour prior to the anticipated reperfusion event and continued through approximately 1 hour following re-establishment of blood flow through the culprit vessel.

The reduction of reperfusion injury, or infarct size, was estimated using the area under the curve (AUC) of the serum creatine kinase (CK) isoenzyme, as well as using magnetic resonance imaging (MRI) performed on the Day 4±1 and on Day 30±7 (both MRI assessments measured infarct size and the ratio of infarct size to myocardial mass). The analyses of cardiac MRI data were performed for both the primary endpoint population and also in all patients who had adequate Day 4/Day 30 cardiac MRI studies.

After completion of the percutaneous coronary intervention (PCI) and stenting, patients received standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and <85 years
* The patient presents with first-time acute, anterior wall STEMI scheduled to undergo primary PCI and stenting.
* The patient has symptoms of cardiac ischemia of ≥10 minutes.
* The patient must demonstrate an anterior wall STEMI with >0.1 millivolt (mV) ST-segment elevation in at least two contiguous precordial leads (i.e., V1-V4) or presumed new left bundle branch block.
* The time from onset of symptoms of cardiac ischemia to the anticipated time of initial PCI balloon inflation does not exceed four (4) hours and it is anticipated that the door-to-balloon time will be <2 hours.
* For female patients of child-bearing potential, an adequate form of contraception must be adhered to prior to entry into the study and for a further 3 months after the follow-up visit. Female patients of childbearing potential must have a negative serum pregnancy test prior to entry into the study.
* Female patients not of childbearing potential (i.e. female patients who are postmenopausal since last regular menses, or have been surgically sterilized at least 1 year prior to screening visit) are eligible to enter the study.
* For male patients with female partners of child-bearing potential, an adequate form of contraception must be adhered to prior to entry into the study and for a further 3 months after the post-study medical.
* Written informed consent obtained that strictly adheres to the written guidelines from the local Institutional Review Board (IRB)/ Ethical Committee (EC).

Exclusion Criteria

* Cardiogenic shock or maximal systolic blood pressure (BP) <80 mm Hg after fluid and/or vasopressor resuscitation on at least two consecutive readings.
* Ongoing vasopressor support.
* Uncontrolled hypertension defined as a systolic BP >180 mm Hg or a diastolic BP >110 mm Hg on at least two consecutive readings.
* Cardiac arrest or arrhythmia requiring prolonged (>5 minutes) chest compressions/ cardiopulmonary resuscitation (CPR).
* Prior coronary artery bypass graft surgery (CABG).
* Prior myocardial infarction (MI).
* Implantable cardioverter-defibrillator (ICD) or permanent pacemaker (PPM) unless known to be MRI safe. The presence of an MRI-compatible pacemaker or other MRI-compatible hardware will not be a contraindication to participation in this trial.
* Known left ventricular ejection fraction <30% prior to the qualifying infarct.
* History of clinically significant hepatic disturbance or chronic renal impairment at the time of admission.
* Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the last 30 days.
* Any known disorder that is associated with immunologic dysfunction (e.g., cancer, lymphoma, a positive serologic test for the human immunodeficiency virus, or hepatitis) more recently than 6 months before presentation or the administration of immunosuppressive drugs within 10 days of the STEMI at doses expected to be associated with immunosuppression including high dose steroids (>2.5 mg/d hydrocortisone or equal potency of synthetic steroids), tumor necrosis factor-alpha (TNF-α) blockers or methotrexate/azathioprine.
* Any condition that, in the Investigator's opinion, would prevent adherence to the requirements of the protocol including language barrier or current alcohol or drug abuse.
* Contraindications (including claustrophobia) to cardiac MRI at study entry.
* Participation in an investigational drug or device study within the 30 days prior to enrollment into the EMBRACE-STEMI Trial or anticipated within the next 4 days.
* Female patients who are pregnant or breastfeeding during the study or intend to within 30 days of receiving study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjan Chakrabarti, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Interventional Cardiology, 185 Pilgrim Rd, Baker 4, Boston, MA 02215; C. M. Gibson, MD, Study Chair — Beth Israel Deaconess Medical Center, Interventional Cardiology, 185 Pilgrim Rd, Baer 4, Boston, MA 02215
Locations (30):
- United States (3):
  - Advanced Medical Research Center, Port Orange, Florida
  - Henry Ford Hospital, Detroit, Michigan
  - Creighton Cardiac Center, Omaha, Nebraska
- Germany (7):
  - Universitätsmedizin Berlin, Charité Campus Benjamin Franklin, Berlin
  - Staedtische Kliniken Bielefeld, Bielefeld
  - Marienhaus Klinikum Eifel, Bitburg
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Herford, Herford
  - Robert-Bosch-Krankenhaus Kardiologie, Stuttgart
  - Helios Klinikum Wuppertal, Herzzentrum Elberfeld, Wuppertal
- Hungary (6):
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Semmelweis Egyetem Kardiológiai Központ, Városmajor u. 68, Budapest
  - Honvédkórház-Állami Egészségügyi Központ, Budapest
  - PTE Klinikai Központ Szívgyógyászati Klinika, Pécs
  - Szent György Kórház, II. Belgyógyászati Osztály, Székesfehérvár
  - Zala Megyei Kórház, Kardiológiai Osztály, Zrínyi Miklós út 1., Zalaegerszeg
- Poland (14):
  - Medical University of Bialystok, Bialystok
  - SPSK Nr 7 Klaskiego Uniwersytetu Medycznego w Katowicach, Gornoslaskie Centrum Medyczne im. Prof. Leszka Gieca, III Oddzial Kardiologii, Zklad Kardiologii Inwazjnejul, Ziolowa 45-47, Katowice
  - SPSK Nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Gornoslaskie Centrum Medyczne im. Prof. Leszaka Gieca, I Oddzial Kardiologii, ul. Ziolowa 45-47, Katowice
  - Wojewodzki Szpital Zespolony w Kielcach, Swietokrzyskie Centrum Kardiologii, Kielce
  - Krakowski Szpital Specjalistyczny im. Jana Pwla II, Centrum Interwencyjnego Leczenia Chorob Serca i Naczyn z Pododdzialem Kariologii Interwencyjnej, Krakow
  - Wojewodzki Specjalistyczny Szpital im WI. Bieganskiego, II Katedra i Klinika Kardiologii Uniwersytetu Medycznego w Lodzi, Pracownia Kardiologii Inwazyinej, ul. Kniaziewicza 1/5, Lodz
  - SP ZOZ Wojewodzkie Centrum Medyczne, Zaklad Diagnostyki Obrazowej, AI. W. Witosa 26, Opole
  - Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii, Oświęcim
  - Szpital Bielanski im. ks. Jerzego Popieluszki, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Pracownia Kardiologii Inwazyjnej, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego, Warsaw
  - Dolnoslaski Szpital Specjalistyczny im. T. Marciniaka, Centrum Medycyny Ratunkowe, Wroclaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Oddzial Kardiologiczny, ul. H. Kamieskiego 73a, Wroclaw
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II w Zamosciu, Oddzial Kardiologii z Pododdzialem Intensywnej Terapil Kardiologicznej, ul. Aleje Jana Pawta II 10, Zamość

REFERENCES:
- [Derived] Daaboul Y, Korjian S, Weaver WD, Kloner RA, Giugliano RP, Carr J, Neal BJ, Chi G, Cochet M, Goodell L, Michalak N, Rusowicz-Orazem L, Alkathery T, Allaham H, Routray S, Szlosek D, Jain P, Gibson CM. Relation of Left Ventricular Mass and Infarct Size in Anterior Wall ST-Segment Elevation Acute Myocardial Infarction (from the EMBRACE STEMI Clinical Trial). Am J Cardiol. 2016 Sep 1;118(5):625-31. doi: 10.1016/j.amjcard.2016.06.025. Epub 2016 Jun 15. PMID 27392509
- [Derived] Chakrabarti AK, Feeney K, Abueg C, Brown DA, Czyz E, Tendera M, Janosi A, Giugliano RP, Kloner RA, Weaver WD, Bode C, Godlewski J, Merkely B, Gibson CM. Rationale and design of the EMBRACE STEMI study: a phase 2a, randomized, double-blind, placebo-controlled trial to evaluate the safety, tolerability and efficacy of intravenous Bendavia on reperfusion injury in patients treated with standard therapy including primary percutaneous coronary intervention and stenting for ST-segment elevation myocardial infarction. Am Heart J. 2013 Apr;165(4):509-514.e7. doi: 10.1016/j.ahj.2012.12.008. Epub 2013 Feb 15. PMID 23537966

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendavia™: Participants received Bendavia (MTP-131) as an IV infusion at 0.05 mg/kg/hr at least 15 minutes but no more than 1 hour prior to the anticipated reperfusion event and continued through approximately 1 hour following re-establishment of blood flow through the culprit vessel via primary percutaneous coronary intervention and stenting.
- Placebo: Participants received placebo as an IV infusion at 60 mL/hr at least 15 minutes but no more than 1 hour prior to the anticipated reperfusion event and continued through approximately 1 hour following re-establishment of blood flow through the culprit vessel via primary percutaneous coronary intervention and stenting.
Period: Overall Study
Arm/Group | Bendavia™ | Placebo
Started | 152 | 148
Completed | 120 | 123
Not Completed | 32 | 25
Not completed — Adverse Event | 7 | 2
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 8 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Technical Issues | 1 | 0
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Infarct, comorbidity, Pt refusal of exam | 0 | 3

BASELINE CHARACTERISTICS:
Population: 300 patients were randomized and only 297 were included in the Safety Population, which consists of all patients who took any fraction of study drug using actual treatment received. If patient was randomized to placebo and received elamipretide, patient's actual treatment was recognized as elamipretide (and vice versa).
Groups:
- Total: Total of all reporting groups
Arm/Group | Bendavia™ | Placebo | Total
Number analyzed (Participants) | 150 | 147 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11) | 60.1 (10.6) | 60.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 28 | 73
  Male | 105 | 119 | 224
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 150 | 146 | 296
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Serum Creatine Kinase Isoenzyme Type Muscle-brain (CK-MB)
Description: Infarct size as measured by the AUC of serum CK-MB at 24 and 72 hours post-PCI
Time Frame: The initial 24 and 72 hours post-percutaneous coronary intervention (PCI)
Population: All participants in the Primary Analysis Population (PAP) for whom CK-MB over the initial 72 hours post-PCI was measured.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 57 | 60
ng*hr/mL
  72 Hours | 6582.0 (3270.6) | 6738.3 (3775.4)
  24 Hours | 5252.2 (2667.9) | 5471.9 (3270.7)

2. Secondary Outcome: AUC of Troponin 1 Enzyme
Description: Infarct size as calculated by the AUC of Troponin I Enzyme over the initial 24 and 72 hours post-PCI
Time Frame: Initial 24 and 72 hours post-PCI
Population: All participants in the Primary Analysis Population (PAP) for whom Troponin 1 Enzyme over the initial 72 hours post-PCI was measured.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 57 | 60
ng*hr/mL
  72 Hours | 5422.9 (3430.9) | 4647.2 (2834.7)
  24 Hours | 3301.4 (2192.9) | 2850.4 (1640.6)

3. Secondary Outcome: Ratio of Volume of Infarcted Myocardium to Left Ventricular Mass
Description: Cardiac infarct size calculated as the ratio of volume of infarcted myocardium to left ventricular mass at Day 30 as measured by MRI.
Time Frame: Day 30 + 7
Population: All participants in the Primary Analysis Population (PAP) for whom ratio of volume of infarcted myocardium and left ventricular mass was measured.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 46 | 47
ratio | 242.3 (87.3) | 225.2 (90.70)

4. Secondary Outcome: Thrombosis in Myocardial Infarction (TIMI) Perfusion Grade Flow at Completion of PCI
Description: TIMI perfusion grade flow at completion of PCI will be categorized as 0,1, or 1.5, 2 or 2.5, 3, and treated as ordinal data, where higher score means better perfusion and lower score means worse perfusion and worse outcome.
Time Frame: Initiation to Completion of PCI, no longer than 4 hours
Population: All participants in the Primary Analysis Population (PAP) for whom Thrombosis in Myocardial Infarction (TIMI) Perfusion Grade Flow at Completion of PCI was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants
  Flow Grade 0 | 0 | 0
  Flow Grade 1 or 1.5 | 0 | 0
  Flow Grade 2 or 2.5 | 6 | 7
  Flow Grade 3 | 52 | 53

5. Secondary Outcome: Corrected TIMI Frame Count
Description: Corrected TIMI Frame Count at Completion of PCI as captured by angiogram and analyzed as a continuous variable.
Time Frame: Completion of PCI, no longer than 4 hours
Population: All participants in the Primary Analysis Population (PAP) for whom corrected TIMI perfusion grade at completion of PCI was measured.
Measure: Mean (Standard Deviation); unit: corrected frame count
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 59
corrected frame count | 79.7 (122.8) | 166.0 (286.8)

6. Secondary Outcome: ST-Segmented Elevation From Pre-PCI to 24 Hours Post-PCI and Presence of ST-Segmented Resolution
Description: ST-Segmented Elevation from pre-PCI to 24 hours post-PCI and Presence of ST-Segmented Resolution by ECG
Time Frame: pre-PCI to 24 hours post-PCI
Population: All participants in the Primary Analysis Population (PAP) for whom the amount of ST-segment elevation resolution from the pre-PCI electrocardiogram to the 24-hour post-PCI ECG was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 56 | 57
Participants
  Complete (>=70% resolution) | 30 | 29
  Partial (<70% resolution) | 22 | 21
  None (<30% resolution) | 4 | 7

7. Secondary Outcome: Change in Serum Creatinine From Baseline
Description: Change in serum creatinine, from baseline (prior to study drug administration) to Day 30 +7 post-PCI
Time Frame: Day 30 +7
Population: All participants in the Primary Analysis Population (PAP) for whom Serum Creatinine was recorded at baseline and Day 30 +7.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
umol/L | 10.55 (17.642) | 88.04 (22.462)

8. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline
Description: Change in eGFR from baseline (prior to study drug administration) to Day 30 +7 post-PCI
Time Frame: Day 30 +/- 7
Population: All participants in the Primary Analysis Population (PAP) for whom Change in eGFR, from baseline to Day 30 +7 was measured.
Measure: Mean (Standard Deviation); unit: mL/min/SSA
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 51 | 50
mL/min/SSA | -12.33 (18.873) | -8.94 (14.242)

9. Secondary Outcome: Cystatin C Change From Baseline
Description: Change in Cystatin C from baseline (prior to study drug administration) to Day 30 +7 post-PCI
Time Frame: Day 30 + 7
Population: All participants in the Primary Analysis Population (PAP) for whom Cystatin C was measured at baseline and Day 30 +7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 53 | 49
mg/L | 0.19 (0.341) | 0.19 (0.226)

10. Secondary Outcome: Blood Urea Nitrogen (BUN) Change From Baseline
Description: Blood Urea Nitrogen (BUN) Change from baseline (prior to study drug administration) to Day 30 + 7 post-PCI
Time Frame: Baseline to Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom BUN at baseline and Day 30 was measured
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 53 | 51
mmol/L | -0.13 (1.603) | 0.13 (2.207)

11. Secondary Outcome: Number and Percent of Grade 1 Episode of Contrast-Induced Nephropathy Post-PCI
Description: Number of Participants with Grade 1 Episode of Contrast-Induced Nephropathy within 48 hours of initial PCI or MRI, based on lab data.
Time Frame: Baseline to 48 hours post PCI or MRI
Population: All participants in the Primary Analysis Population (PAP) for whom Contrast-Induced Nephropathy within 48 hours of initial PCI or MRI, based on lab data, was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants
  Yes | 17 | 11
  No | 41 | 49

12. Secondary Outcome: Immediate Myocardial Complications: Ventricular Tachycardia or Fibrillation
Description: Number and percent of participants with Immediate Myocardial Complications: Ventricular Tachycardia or Fibrillation Requiring Medical Intervention
Time Frame: Baseline up to 1 hour post-PCI
Population: All participants in the Primary Analysis Population (PAP) for whom Immediate Myocardial Complications--Ventricular Tachycardia or Fibrillation Requiring Medical Intervention--was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants
  Yes | 2 | 3
  No | 56 | 57

13. Secondary Outcome: Immediate Myocardial Complications: Mechanical Complications
Description: Number and Percent of Participants with Immediate Myocardial Complications: Mechanical Complications: (Free wall Rupture, Ventricular Septal Defect, Ischemic Mitral Regurgitation)
Time Frame: Baseline up to 1 hour post-PCI
Population: All participants in the Primary Analysis Population (PAP) for whom immediate Myocardial Complications (Mechanical Complications: Free wall Rupture, Ventricular Septal Defect, Ischemic Mitral Regurgitation) was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants | 1 | 0

14. Secondary Outcome: Emergency Use of Medications During PCI Procedure
Description: Emergency Use of Nitroprusside, Calcium Channel Blocker, Adenosine Administration During the PCI Procedure
Time Frame: Initiation to Completion of PCI, no longer than 4 hours
Population: All participants in the Primary Analysis Population (PAP) for whom Emergency Use of Nitroprusside, Calcium Channel Blocker, or Adenosine Administration During the PCI Procedure) was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants
  Yes | 5 | 3
  No | 53 | 57

15. Secondary Outcome: ProB-type Natriuretic Peptide (NT-proBNP) Change From Baseline to Day 30
Description: NT-proBNP: Change from baseline to Day 30 +7 (Laboratory marker for chronic heart failure (CHF) and systemic inflammation.)
Time Frame: Baseline to Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom NT-proBNP had been measured at baseline and Day 30 +7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 51 | 51
pg/mL | 1828.45 (3427.408) | 1582.67 (1502.985)

16. Secondary Outcome: High Sensitivity C-Reactive Protein (hsCRP): Change From Baseline to Day 30
Description: High Sensitivity C-Reactive Protein (hsCRP): Change from baseline to Day 30 +7 (Laboratory Marker for CHF and Systemic Inflammation)
Time Frame: Baseline to Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom hsCRP was measured at baseline and Day 30.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 51 | 45
mg/L | -1.03 (7.072) | -0.91 (7.024)

17. Secondary Outcome: Left Ventricular (LV) Ejection Fraction (%)
Description: Difference in Left Ventricular (LV) Ejection Fraction (%) from Day 4 To Day 30
Time Frame: Day 4 to Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom LV ejection fraction was measured at Day 4 and Day 30
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 47 | 53
percentage of blood volume | 2.1 (6.4) | 2.5 (8.3)

18. Secondary Outcome: Difference Between Left Ventricular End Diastolic Volume, Corrected
Description: Difference between Left Ventricular End Diastolic Volume Corrected for Body Surface Area between Day 4 and Day 30
Time Frame: Day 4 and Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom Left Ventricular End Diastolic Volume Corrected for Body Surface Area was measured on Day 4 and Day 30
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 45 | 52
mL/m2 | 8.6 (12.6) | 6.2 (15.1)

19. Secondary Outcome: Difference Between Left Ventricular End Systolic Volume, Corrected
Description: Difference between Left Ventricular End Systolic Volume Corrected for Body Surface Area from Day 4 and Day 30
Time Frame: Day 4 and Day 30
Population: All participants in the Primary Analysis Population (PAP) for whom Left Ventricular End Systolic Volume was measured at Day 4 and Day 30
Measure: Mean (Standard Deviation); unit: mL/m²
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 45 | 52
mL/m² | 2.7 (8.0) | 1.5 (12.5)

20. Secondary Outcome: Chronic Heart Failure
Description: Number and Percentage of Patients with Clinical Events: Chronic Heart Failure beginning within 24 hours after PCI but within the duration of the index hospitalization (Subjects with CHF started within 24 hours after the last balloon deflation while the patient was still in the hospital {including patients who had missing discharge date}).
Time Frame: Within 24 hours after PCI
Population: All participants in the Primary Analysis Population (PAP) for whom CHF which began within 24 hours after PCI but within the duration of the index hospitalization was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendavia™ | Placebo
Number analyzed (Participants) | 58 | 60
Participants
  Yes | 8 | 15
  No | 50 | 45

ADVERSE EVENTS:
Arm/Group | Bendavia™ | Placebo
All-Cause Mortality (participants affected / at risk) | 10/150 | 3/147
Serious Adverse Events (participants affected / at risk) | 20/150 | 14/147
Other Adverse Events (participants affected / at risk) | 112/150 | 106/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendavia™ (N=150) | Placebo (N=147)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 2
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 4 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 1
Femoral Artery Embolism (Vascular disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Sudden Cardiac Death (General disorders) | 1 | 0
Thrombosis in Device (General disorders) | 2 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternum Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1 — asystolia
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatic Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrioventricular Block (Cardiac disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Ischemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Intracardiac Thrombus (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendavia™ (N=150) | Placebo (N=147)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 9 | 14
Claustrophobia (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 7 | 1
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 6 | 2
Hypotonia (Nervous system disorders) | 3 | 3
Syncope (Nervous system disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Urinary tract infection (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 3 | 4
Pyrexia (General disorders) | 5 | 9
Non-cardiac chest pain (General disorders) | 9 | 5
Catheter site pain (General disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 8 | 7
Nausea (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Constipation (Gastrointestinal disorders) | 1 | 4
Blood potassium decreased (Investigations) | 2 | 3
Ejection fraction decreased (Investigations) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Angina Pectoris (Cardiac disorders) | 11 | 6
Atrial Fibrillation (Cardiac disorders) | 6 | 8
Bradycardia (Cardiac disorders) | 0 | 3
Cardiac Failure (Cardiac disorders) | 28 | 29
Cardiac Failure Congestive (Cardiac disorders) | 5 | 5
Coronary Artery Disease (Cardiac disorders) | 5 | 5
Coronary Artery Stenosis (Cardiac disorders) | 3 | 4
Intracardiac Thrombus (Cardiac disorders) | 9 | 10
Mitral Valve Incompetence (Cardiac disorders) | 3 | 1
Pericardial effusion (Cardiac disorders) | 0 | 3
Ventricular extrasystoles (Cardiac disorders) | 4 | 1
Ventricular Tachycardia (Cardiac disorders) | 4 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 12 | 7
Glucose Tolerance Impairment (Metabolism and nutrition disorders) | 5 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 30 | 19
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 27
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Type 2 Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 3
Haematoma (Vascular disorders) | 4 | 4
Hypertension (Vascular disorders) | 11 | 9
Hypotension (Vascular disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes